CLINICAL TRIAL: NCT00623636
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Phase 3 Study of MAP0004 in Adult Migraineurs for a Single Migraine Followed by Open Label Extension.
Brief Title: Phase 3 Study of MAP0004 in Adult Migraineurs
Acronym: FREEDOM301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP0004 CL P301
Record Dates: First submitted 2008-02-07; First posted 2008-02-26 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Migraine Disorders
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAP0004 (Experimental): MAP0004 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat qualifying migraines for up to an additional 52 weeks.
  Interventions: Drug: MAP0004
- Placebo (Other): Placebo 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat qualifying migraines for up to 52 weeks.
  Interventions: Drug: MAP0004; Drug: Placebo

INTERVENTIONS:
Drug: MAP0004 — MAP0004 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat qualifying migraines for up to an additional 52 weeks. Placebo treated patients will receive MAP0004 1.0mg inhaled to treat qualifying migraines for up to 52 weeks only.
Drug: Placebo — Placebo 1.0mg inhaled to treat a qualifying migraine up to 8 weeks.
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel group study of MAP0004 in adult migraineurs. Subjects will self administer study drug in the outpatient setting.

ELIGIBILITY:
Major Inclusion Criteria:

* Male or female between 18 and 65 years of age.
* History of episodic, acute migraine (with or without aura) with onset prior to 50

Major Exclusion Criteria:

* Known allergy or sensitivity or contraindication to study drugs or their formulations
* History of chronic pulmonary disease, coronary artery disease (CAD), liver disease, kidney disease, seizures, stroke, or major psychiatric condition.
* Any condition that, in the opinion of the Investigator, would make the subject unsuitable for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MAP Pharmaceuticals a Wholly Owned Subsidiary of Allergan
Locations (1):
- Swedish Pain and Headache Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Tepper SJ, Kori SH, Borland SW, Wang MH, Hu B, Mathew NT, Silberstein SD. Efficacy and safety of MAP0004, orally inhaled DHE in treating migraines with and without allodynia. Headache. 2012 Jan;52(1):37-47. doi: 10.1111/j.1526-4610.2011.02041.x. Epub 2011 Nov 22. PMID 22106843
- [Derived] Tepper SJ, Kori SH, Goadsby PJ, Winner PK, Wang MH, Silberstein SD, Cutrer FM. MAP0004, orally inhaled dihydroergotamine for acute treatment of migraine: efficacy of early and late treatments. Mayo Clin Proc. 2011 Oct;86(10):948-55. doi: 10.4065/mcp.2011.0093. PMID 21964172
- [Derived] Aurora SK, Silberstein SD, Kori SH, Tepper SJ, Borland SW, Wang M, Dodick DW. MAP0004, orally inhaled DHE: a randomized, controlled study in the acute treatment of migraine. Headache. 2011 Apr;51(4):507-17. doi: 10.1111/j.1526-4610.2011.01869.x. PMID 21457235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a Double-blind period for 8 weeks followed by an open-label period that lasted an additional 52 weeks. All patients participating in the open-label period received MAP0004.
Groups:
- Placebo: Placebo 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat a qualifying migraine for up to an additional 52 weeks.
Period: Double Blind
Arm/Group | Placebo | MAP0004
Started | 452 | 450
Completed | 419 | 422
Not Completed | 33 | 28
Period: Open Label
Arm/Group | Placebo | MAP0004
Started | 0 (Eligible double-blind placebo patients received MAP0004 in the open-label period.) | 675 (Includes eligible Placebo and MAP0004 patients from the double-blind period.)
Completed | 0 | 263
Not Completed | 0 | 412

BASELINE CHARACTERISTICS:
Population: mITT population was defined as all randomized subjects who reported a qualifying migraine and received at least one dose of study treatment, and had at least one post-treatment efficacy evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MAP0004 | Total
Number analyzed (Participants) | 397 | 397 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (11.67) | 40.5 (11.30) | 40.1 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362 | 365 | 727
  Male | 35 | 32 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Pain Relief at 2 Hours From Time of First Dose
Description: Pain relief at 2 hours was defined as change in rating from severe or moderate (score 3 or 2) to a rating of none or mild (score 0 or 1) at the 2-hour time point and no usage of rescue medications from the time of first dose to 2 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 136 | 231

2. Primary Outcome: Number of Subjects Photophobia Free at 2 Hours From Time of First Dose
Description: Photophobia free at 2 hours was defined as a rating of none (score 0) at the 2-hour time point and no usage of rescue medications from the time of first dose to 2 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 107 | 182

3. Primary Outcome: Number of Subjects Phonophobia Free at 2 Hours From Time of First Dose
Description: Phonophobia free at 2 hours was defined as a rating of none (score 0) at the 2-hour time point and no usage of rescue medications from the time of first dose to 2 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 133 | 208

4. Primary Outcome: Number of Subjects Nausea Free at 2 Hours From Time of First Dose
Description: Nausea free was defined as a rating of none (score 0) at the 2-hour time point and no usage of rescue medications from the time of first dose to 2 hours post-dose.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 234 | 266

5. Secondary Outcome: Number of Subjects With Sustained Pain Relief From 2 to 24 Hours
Description: Sustained Pain Relief was defined as a rating of none or mild (score 0 or 1) at the 2-hour time point that was maintained during the 2-24 hour post-dose period and no use of rescue medication from the time of first dose to 24 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: From 2 to 24 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 76 | 166

6. Secondary Outcome: Number of Subjects Whose Time to Pain Relief Occurred Within 2 Hours
Description: The number of subjects who reported pain relief (score of 0 or 1) at any time within the 2 hours following the time of first dose and who did not use rescue medication on or prior to this point. Subjects who did not reach pain relief by the end of the time period were not included.
  The 4-point scale from the International Headache Society was used: 0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from the first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 156 | 244

7. Secondary Outcome: Number of Subjects With Pain Relief at 4 Hours
Description: Pain Relief at 4 hours was defined as a change in rating from severe or moderate (score 3 or 2) to none or mild (score 0 or 1) at the 4-hour time point and no use of rescue medication from the time of first dose to 4 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 4 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 145 | 254

8. Secondary Outcome: Number of Subjects With Pain Relief at 10 Minutes
Description: Pain Relief at 10 minutes was defined as a change in rating from severe or moderate (score 3 or 2) to none or mild (score 0 or 1) at the 10 minute time point and no use of rescue medication from the time of first dose to 2 hours.
  The 4-point scale from the International Headache Society was used:
  0 = none; 1 = mild symptom, not interfering with normal daily activities; 2 = moderate symptom, causing some restriction to normal activities; 3 = severe, leading to inability to perform daily activities
Time Frame: 2 hours from time of first dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MAP0004
Number analyzed (Participants) | 397 | 397
participants | 30 | 37

ADVERSE EVENTS:
Description: All subjects who received any dose of study treatment in the double-blind or open-label study period and had at least one post-dose safety evaluation were included in the adverse events analysis.
Groups:
- Double-blind Placebo: Placebo 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat a qualifying migraine for up to an additional 52 weeks.
- Double-blind MAP0004: MAP0004 1.0mg inhaled to treat a qualifying migraine up to 8 weeks followed by MAP0004 1.0mg inhaled to treat qualifying migraines for up to an additional 52 weeks.
- Open-label MAP0004: MAP0004 1.0mg inhaled to treat a qualifying migraine for up to an additional 52 weeks.
Arm/Group | Double-blind Placebo | Double-blind MAP0004 | Open-label MAP0004
Serious Adverse Events (participants affected / at risk) | 0/404 | 0/410 | 14/638
Other Adverse Events (participants affected / at risk) | 60/404 | 86/410 | 454/638
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=404) | Double-blind MAP0004 (N=410) | Open-label MAP0004 (N=638)
Aplastic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Decompression sickness (Injury, poisoning and procedural complications) | 0 | 0 | 1
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=404) | Double-blind MAP0004 (N=410) | Open-label MAP0004 (N=638)
Pharmaceutical Product Compaint (Social circumstances) | 11 | 25 | 51 — Medication Aftertaste
Nausea (Gastrointestinal disorders) | 7 | 18 | 78
Vomiting (Gastrointestinal disorders) | 3 | 8 | 33
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 11 | 93
Sinusitis (Infections and infestations) | 5 | 3 | 65
Nasopharyngitis (Infections and infestations) | 15 | 8 | 67
Influenza (Infections and infestations) | 0 | 3 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.